CLINICAL TRIAL: NCT06541288
Title: A Prospective Cohort Study Comparing Artificial Intelligence Multimodal Fusion Prediction Models With Conventional Imaging Assessment for the Diagnosis of Pelvic Lymph Node Metastasis in Cervical Cancer
Brief Title: A Prospective Cohort Study Comparing AI Prediction Model With Imaging Assessment to Diagnose Lymph Node Metastasis in Cervical Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xin Wu, Deputy Chief of Gynecologic Oncology, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: FUOBGY-2024-64
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI Prediction Model (Experimental)
  Interventions: Diagnostic Test: AI Prediction Model
- Conventional Imageing Assessment (Active Comparator)
  Interventions: Diagnostic Test: Conventional Imageing Assessment

INTERVENTIONS:
Diagnostic Test: AI Prediction Model — Pelvic MRI was performed after pathologic diagnosis clarified the diagnosis of cervical cancer. Further pelvic lymph node metastasis status was determined by artificial intelligence multimodal fusion prediction modeling
  Arms: AI Prediction Model
Diagnostic Test: Conventional Imageing Assessment — Pelvic MRI was performed after pathologic diagnosis clarified the diagnosis of cervical cancer.Further pelvic MRI images are read by a specialized imaging physician to determine pelvic lymph node status.
  Arms: Conventional Imageing Assessment

SUMMARY:
The goal of this prospective cohort study is to learn whether artificial intelligence multimodal fusion prediction models are effective in diagnosing pelvic lymph node metastasis in cervical cancer. The main question it aims to answer is: can artificial intelligence multimodal fusion prediction models improve the accuracy of preoperative diagnosis of pelvic lymph node metastasis in cervical cancer? The researchers compared the AI multimodal fusion prediction model with traditional imaging physician assessments to see if the prediction model could yield more accurate lymph node metastasis determinations. Participants will undergo pelvic MRI after pathologically confirming a diagnosis of cervical cancer, and the results will be used to determine pelvic lymph node metastasis status by the predictive model and the imaging physician, respectively. Subsequent pathology results after surgical lymph node clearance will be used as the gold standard to determine the accuracy of the two preoperative lymph node diagnostic modalities.

ELIGIBILITY:
Inclusion criteria:

1. patients with preoperative diagnosis of invasive cervical cancer stage I-III, with any type of pathology, and patients who underwent radical/modified radical cervical cancer surgery + pelvic lymph node dissection in our hospital or sub-center;
2. Age ≥18 years and ≤80 years;
3. patients who underwent preoperative pelvic MRI (plain/enhanced) imaging in our hospital or sub-centers.

Exclusion criteria:

1. patients during pregnancy or lactation, patients with abortion within 42 days;
2. patients who are undergoing or have undergone preoperative neoadjuvant chemotherapy or radiotherapy for this cervical cancer;
3. Patients with other malignant tumors within 5 years;
4. Combination of other underlying diseases that may lead to enlarged pelvic lymph nodes;
5. patients whose preoperative pelvic MRI date is more than 1 month from the day of surgery;
6. poor quality imaging images that are unrecognizable.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy in determining pelvic lymph node metastasis | The time frame was from subject enrollment until surgical pathology results were obtained. The time between subject enrollment and the availability of surgical pathology results was approximately 1 to 1.5 months.
  After the subjects underwent surgical treatment, surgical pathology served as the gold standard for evaluating the accuracy of the AI predictive model in comparison to traditional imaging diagnosis. In the statistical analysis phase, sensitivity and specificity were utilized as the primary indicators to assess the accuracy of both diagnostic modalities.

CONTACTS AND LOCATIONS:
Locations (1):
- The Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No